CLINICAL TRIAL: NCT03376100
Title: Ultrasound Guided Radial and Median Nerve Blocks Versus Haematoma Block for Closed Reduction of Distal Forearm Fractures; a Randomised Controlled Trial.
Brief Title: Distal Nerve Blocks for Closed Reduction of Distal Forearm Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Regionshospitalet Viborg, Skive (Other)
Collaborators: Aalborg University Hospital (Other); Randers Regional Hospital (Other); Herning Hospital (Other)
Responsible Party: Principal Investigator, Christoffer Grant Sølling, Consultant, Head of Research, MD, PhD, Regionshospitalet Viborg, Skive
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 030021
Record Dates: First submitted 2017-12-06; First posted 2017-12-18 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Fracture Closed of Lower End of Forearm, Unspecified

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Patients with distal forearm fractures randomized to Hematoma Block.
  Interventions: Procedure: Hematoma Block
- Intervention Group (Active Comparator): Patients with distal forearm fractures randomized to Ultrasound guided nerve block
  Interventions: Procedure: Ultrasound guided nerve blocks

INTERVENTIONS:
Procedure: Ultrasound guided nerve blocks — Ultrasound guided nerve blocks of the radial and median nerves
  Arms: Intervention Group
Procedure: Hematoma Block — Conventional local anesthetic method using hematoma block
  Arms: Control Group

SUMMARY:
Randomized controlled trial comparing the standard haematoma block used for reduction of distal forearm fractures in the Emergency Department with ultrasound guided nerveblocks. The investigators hypothesize that ultrasound guided blocking of the radial and median nerves will improve fracture reduction satisfaction for the true Colles' fractures and improve analgesia for reduction of all distal forearm fracture types compared to the standard haematoma block.

DETAILED DESCRIPTION:
Multicenter randomized controlled trial comparing the standard hematoma block as the local anaesthetic procedure for reduction of distal forearm fracture with ultrasound guided radial and median nerve blocks.

Among all dislocated fractures of the distal forearm only the true Colles' fracture can potentially be treated adequately with a closed reduction and a cast, while the other fracture types are unstable by definition and require surgical stabilization. Most dislocated forearm fractures, however, require a primary reduction and this procedure requires the patient to be relieved of pain and the muscle traction on the fracture to be minimal. The conventional local anaesthetic procedure used in Denmark is the hematoma block where the local anaesthetic agent is injected directly in the fracture. This is done using either a blind technique or with the aid of X-ray to visualize the fracture line. The radial and median nerves supply periosteal innervation for the radius and the ulna as well as muscular innervation for the majority of muscles in the forearm and wrist. Blocking these nerves at the level of the cubital fossa should relieve pain and minimize muscular traction when performing closed reductions on distal forearm fractures.

The investigators hypothesize that ultrasound guided blocking of the radial and median nerves will improve fracture reduction satisfaction for the true Colles' fractures and improve analgesia for reduction of all fracture types compared to the standard haematoma block.

Patients eligible for screening for inclusion are identified in the Emergency Department (ED) at all recruitment sites upon primary contact. When an X-ray has revealed the relevant fracture, the ED-staff will call the available anaesthesiologist or anaesthesiologist trainee who will perform the inclusion process and randomisation. Participants will be randomized in either the intervention or the control group using the online randomization tool Research Electronic Data Capture (REDCap, Aarhus University, Denmark). In both groups, the reduction process will begin 10 minutes after the block has been performed. The technique for the actual reduction may vary amongst physicians. To best reflect the clinical practices and to avoid the risk of an insufficient reduction due to the physician being forced to comply to a technique unfamiliar to him, no further standardisation will be made in this regard. Following casting of the fracture a control X-ray will be performed and subsequently evaluated independently by two skilled orthopaedic surgeons to establish if the reduction was satisfactory. In case of disputes a third orthopaedic surgeon will evaluate the X-ray and make a final ruling. The fracture will be deemed satisfactory using a binary outcome measure (yes/no) if all the following requirements set by the National Clinical Guideline for Treatment of Distal Radius Fractures are met.

Binary data, including primary endpoint will be analysed using chi squared test. For normally distributed measurements the differences between groups will be compared using Student´s t-test. Variables considered not to be normally distributed will be analysed by Mann-Whitney´s U-test. Two-tailed P-values < 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion criteria

* Presence of a closed distal forearm fracture in need of a closed reduction
* Age > 18 years
* Legally competent

Exclusion criteria

* Inability to give informed consent
* Allergy or intolerance towards local anaesthetics
* Infection or burns at either injection site
* Multi trauma (defined as other fractures or significant injuries)
* Known pregnancy
* Participation in other studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 268 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-11-13 (Actual); Study Completion 2024-05-20 (Actual)

PRIMARY OUTCOMES:
Reduction satisfaction | Within 8 hours from admission
  Based on objective X-ray measures according to the Danish National Guideline for Treatment of Distal Forearm Fractures. The primary outcome applies for the true Colles' fractures only.

SECONDARY OUTCOMES:
Pain, during reduction | Within 8 hours from admission
  Pain score using an 11-step numeric rating scale (0-1-2-3-4-5-6-7-8-9-10, with 0 being no pain and 10 being worst pain imanigable)
Pain, when local anaesthetic is injected | Within 8 hours from admission
  Pain score using an 11-step numeric rating scale (0-1-2-3-4-5-6-7-8-9-10, with 0 being no pain and 10 being worst pain imanigable)
Time spent on reduction | Within 8 hours from admission
  Time stamp start; when reduction begins. Time stamp end; when casting is complete
Secondary fracture dislocation | Records obtained 2 months after primary treatment
  Measured by the need for surgical stabilization

CONTACTS AND LOCATIONS:
Overall Officials: Anette B Christensen, MD, Principal Investigator — Dept. Anesthesiology-Intensive Care Medicine, Reional Hospital Viborg
Locations (1):
- Dept. Anesthesia and Intensive Care, Viborg Regional Hospital, Viborg, Denmark

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-11-02): https://cdn.clinicaltrials.gov/large-docs/00/NCT03376100/Prot_SAP_001.pdf
  • Informed Consent Form (2017-12-05): https://cdn.clinicaltrials.gov/large-docs/00/NCT03376100/ICF_000.pdf